CLINICAL TRIAL: NCT00715182
Title: A Phase I/II Multi-center, Open Label Study of TKI258 Administered Orally on an Intermittent Schedule in Adult Patients With Advanced or Metastatic Renal Cell Cancer (RCC)
Brief Title: A Phase I/II Study to Assess the Safety and Efficacy of TKI258 for the Treatment of Refractory Advanced/Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2107; 2007-004391-39 (EudraCT Number)
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2013-01

CONDITIONS: Advanced/ Metastatic Renal Cell Cancer
Keywords: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (1):
- TKI258 (Experimental)
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258

SUMMARY:
This is a phase I/II open-label study to delineate the safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of TKI258. The eligible subject population consists of subjects who have been diagnosed with advanced or metastatic renal cell cancer that is refractory to standard therapy or for which no curative standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* For phase I, confirmed advanced/ metastatic renal cell carcinoma for which no other therapeutic options exist.
* For phase II, must have been previously treated with VEGF receptor tyrosine kinase inhibitor (sunitinib and/or sorafenib).
* For phase II, must have at least one measurable lesion at baseline.
* For both phase I & II, measurable histologically or cytology confirmed progressive metastatic renal cell carcinoma with predominant clear cell histology (>50%).
* At least 4 weeks must have elapsed since any prior anti-cancer therapy (6 weeks for nitrosoureas or mitomycin C).
* Must have recovered from adverse events (to grade 1 or less toxicity according to CTCAE 3.0) due to agents administered more than 28 days earlier.
* Must be eighteen years of age or older
* ECOG performance status 0 or 1.
* Must meet baseline laboratory requirement
* Life expectancy greater than or equal to 12 weeks.
* Signed and witnessed informed consent prior to any screening procedures.

Exclusion Criteria:

* Concurrent therapy with any other investigational agent within 28 days prior to baseline.
* Pregnant or breast feeding women.
* Clinically significant cardiac disease (New York Heart Association, Class III or IV) or impaired cardiac function or clinically significant cardiac diseases.
* Uncontrolled infection.
* Diabetes mellitus with signs of clinically significant peripheral vascular disease.
* Previous pericarditis; clinically significant pleural effusion in the previous 12 months or current ascites requiring two or more interventions/month.
* Known pre-existing clinically significant disorder of the hypothalamic-pituitary axis, adrenal or thyroid glands.
* Prior acute or chronic pancreatitis of any etiology.
* Acute and chronic liver disease and all chronic liver impairment.
* Malabsorption syndrome or uncontrolled gastrointestinal symptoms (such as nausea, diarrhea and vomiting) with toxicity greater than NCI CTCAE grade 2.
* Other severe, acutem or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results and, in the judgement of the investigator, would make the subject inappropriate for this study.
* Treatment with any of the medications that have a potential risk of prolonging the QT interval or inducing Torsades de Points and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* Use of ketoconazole, erythromycin, carbamazapine, phenobarbital, rifampin, phenytoin and quinidine 2 weeks prior to baseline.
* Major surgery within 28 days prior to starting study drug or who have not recovered from side effects of such therapy.
* Known diagnosis of HIV infection (HIV testing is not mandatory).
* History of another clinically significant primary malignancy that requires active intervention.
* Patients with brain metastases as assessed by radiologic imaging.
* Alcohol or substance abuse disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Phase I: To determine the MTD of TKI258, administered orally on a 5 days on/2 days off schedule to adult patients with advanced or metastatic RCC whose diseases have progressed despite standard therapy or for whom no standard anticancer therapy exists. | at end of phase I
Phase II: To determine anti-tumor activity of TKI258 in advanced or metastatic RCC patients with predominant clear cell histology that have been previously treated with VEGF receptor tyrosine kinase inhibitor (sunitinib and/or sorafenib). | at end of phase II

SECONDARY OUTCOMES:
To assess the safety profile of TKI258 | cycle 1: day 1,8,15,26; cycle 2: day 15, 28; cycle 3+: day 28 & at end of study
To assess the effect of TKI258 on plasma biomarkers, pre- and post-treatment | cycle 1: day 1,15,26; cycle 2: 15 & 28; every other cycles: day 28 & at end of study
To explore the pharmacokinetic and pharmacodynamic relationship | end of study
To characterize the single and multiple-dose PK profiles of oral TKI258 | cycle 1: day 1, 8, 15 &26; cycle 2 & 3: day 15 & 28
Progression free survival and over all survival | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (3):
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Seattle, Washington
- France (2):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, München
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Madrid, Spain
- Taiwan (3):
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei

REFERENCES:
- See also: Results for CTKI258A2107 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9363